CLINICAL TRIAL: NCT00004694
Title: Study of Heparin Prophylaxis of Hereditary Angioedema Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 199/13356; UI-9311397; UI-FDR001001
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-04

CONDITIONS: Angioedema
Keywords: genetic diseases and dysmorphic syndromes; hereditary angioedema; rare disease
MeSH Terms: conditions — Angioedema; Genetic Diseases, Inborn; Angioedemas, Hereditary; Rare Diseases | interventions — Heparin

INTERVENTIONS:
Drug: heparin

SUMMARY:
OBJECTIVES:

I. Determine the safety and efficacy of inhaled and subcutaneously administered heparin in the treatment of hereditary angioedema.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, 3 way crossover study.

All patients complete diary cards for the first month of the study in order to determine compliance in providing a daily record of symptoms and medication taken. All compliant patients receive subcutaneously injected heparin twice daily, inhaled heparin daily, or matched saline placebo in a random order. Each of the three drug administration periods lasts 2 months, for a total of 6 months of treatment. Patients who have a flare in disease activity that requires hospitalization are terminated from that drug administration period of the study.

Patients are followed biweekly during the first month and again at the end of the second month for each of the three 2 month drug administration periods.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Confirmed diagnosis of hereditary angioedema (HAE) based upon C4 antigenic level, positive family history, and C1 inhibitor (C1INH) antigenic level (Type I HAE) or functional level (Type II HAE)
* Functional C1 within normal levels if diagnosis of acquired C1INH is possible
* Negative family history will not exclude as long as patient meets all other criteria, has normal C1 level, and has no evidence of acquired C1INH deficiency
* History of symptoms of HAE including episodic swelling, abdominal pain, and/or respiratory difficulty
* Experiencing a minimum of 1-2 HAE episodes within 6 weeks

--Prior/Concurrent Therapy--

* Endocrine therapy: Anabolic steroids allowed as long as dose has not been changed in at least 30 days
* Other: No concurrent and at least 1 week since prior aspirin, nonsteroidal antiinflammatory agents, dipyridamole, Coumadin-like drugs, or any other medication having an effect on coagulation or platelets

--Patient Characteristics--

* Hematopoietic: No clinically significant history of hematologic disease
* Hepatic: No clinically significant history of hepatic disease
* Renal: No clinically significant history of renal disease
* Cardiovascular: No clinically significant history of cardiac disease or hypertension
* Pulmonary: No clinically significant history of pulmonary disease
* Other: No contraindication to the use of inhaled or subcutaneous heparin No drug allergy that would interfere with the study No clinically significant history of: Malignancy Diabetes mellitus Neurologic disease Immunologic disease Bleeding disorder Infirmity No history of drug abuse, alcoholism, psychosis, or other psychological/psychiatric disorder

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 1994-01; Study Completion 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: John M. Weiler, Study Chair — University of Iowa